CLINICAL TRIAL: NCT06239493
Title: IVUS-Guided Treatment for Percutaneous Vascular Interventions
Acronym: IGT-PVI
Status: Suspended | Type: Observational
Why Stopped: Business Decision
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: 200421
Record Dates: First submitted 2023-12-18; First posted 2024-02-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: CAD; PAD; DVT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- IVUS GUIDED: Those undergoing an already planned IVUS guided treatment for percutaneous vascular interventions
  Interventions: Diagnostic Test: IVUS Guided

INTERVENTIONS:
Diagnostic Test: IVUS Guided — Those already undergoing an IVUS guided percutaneous vascular intervention

SUMMARY:
The main objective of the study is to survey and improve the IVUS image quality and X-ray system interoperability by collecting Procedural Data (e.g. raw, pre- processed ultrasound and X-ray data, endpoints such as fluoroscopy time, contrast load and radiation dose, workflow details) during routine intravascular procedures to assure adherence to the high standards of quality during care delivery and promote procedural standardization.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm study to collect procedural data (e.g., raw, pre-processed IVUS, X-ray, and other procedural data) for image quality, workflow and interoperability assessments. Example of additional procedural endpoint data (e.g., time for fluoroscopy and IVUS, contrast load and radiation dose, workflow details, etc.) will be collected. The study will be conducted in a phased approach.

Since the collection of IVUS raw data with a second non-diagnostic pullback affects procedure time, the two aspects of this study - collection of raw IVUS data and procedural data, will be separated until IVUS raw data can be collected directly from the IVUS system with no additional procedural time.

ELIGIBILITY:
Inclusion Criteria:

1. The Patient is ≥18 years of age.
2. Patient is scheduled to undergo percutaneous vascular intervention - peripheral vascular or coronary PCI procedure.

Exclusion Criteria:

1. Patients not meeting the instructions for use (IFU) of the respective IVUS catheters.
2. Patients with lesions or vessel segments deemed unsafe for multiple IVUS pullbacks.
3. Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All comers aged 18 and older scheduled to undergo a percutaneous vascular intervention.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Improve | Procedure (one visit)
  Analyze IVUS images for improvement using manual and automated visualization

SECONDARY OUTCOMES:
Procedural IVUS TIME | Procedure (one visit)
  Procedural time will be recorded. IVUS time of insert and time of removal
PROCEDURAL RADIATION DOSE | Procedure (one visit)
  Radiation dose used during procedure will be recorded
PROCEDURAL AMOUNT OF CONTRAST USED | Procedure (one visit)
  Amount of contrast used during procedure will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Eric Secemsky, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (5):
- United States (5):
  - Southwest Cardiovascular Associates, Mesa, Arizona
  - Pulse Cardiovascular, Scottsdale, Arizona
  - Center for Advanced Cardiac and Vascular Interventions, Tarzana, California
  - Pacific Cardiovascular and Vein Institute, Ventura, California
  - Community Healthcare System, Munster, Indiana

IPD SHARING:
Plan to Share IPD: Undecided